CLINICAL TRIAL: NCT05436730
Title: The Role of Ambulatory Blood Pressure Characteristics, Features of the Structural and Functional Vascular Wall State, the Presence and Severity of Obstructive Sleep Apnea Syndrome in Predicting the "Escape" Phenomenon of the Antihypertensive Therapy Efficacy.
Brief Title: "Escape" Phenomenon of the Antihypertensive Therapy Efficacy
Acronym: ESCAPE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Federal State Budgetary Institution NATIONAL MEDICAL RESEARCH CENTRE OF CARDIOLOGY NAMED AFTER ACADE (Other Government)
Responsible Party: Principal Investigator, Mikhailova Oksana, Dr., clinical reseacher, National Medical Research Center for Cardiology, Ministry of Health of Russian Federation
Other Study IDs: 115061870017
Record Dates: First submitted 2022-06-22; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Arterial Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- "Escape" Phenomenon of the Antihypertensive Therapy Efficacy: Men and women aged 18-90 years with arterial hypertension grade 1-3, stage I-II and initially achieved target BP levels while taking 2-3-component AHT.
  Interventions: Device: Ambulatory blood pressure measurement device; Device: Sphygmocor; Device: VaSera-VS; Device: Somnocheck

INTERVENTIONS:
Device: Ambulatory blood pressure measurement device — Assessment of the 24-h blood pressure profile
  Other Names: BpLab
Device: Sphygmocor — Assessment of the arterial stiffness
Device: VaSera-VS — Assessment of the arterial stiffness
Device: Somnocheck — Assessment of the sleep breath disturbances

SUMMARY:
A little attention is paid to the AHT efficacy escaping problem, which can be explained by the AHT correction simplicity and rapid achievement of the target BP level. Nevertheless, modern statistic data on the effective AH treatment described above let us assume that AHT correction is either totally absent or is untimely in case of the "escape" phenomenon development. This could be one of the main reasons for the high prevalence of ineffective AH treatment. The aim of this study is to determine AHT efficacy "escape" phenomenon timeline and its predictors in hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* Arterial hypertension (AH) grade 1-3, stage I-II
* High compliance during the follow-up period (≥ 85%)
* Initially achieved target office BP levels while taking 2-3-component AHT

Exclusion Criteria:

* Secondary AH
* Resistant AH,
* AH III stage,
* PAP- therapy,
* type 2 diabetes mellitus,
* pregnancy
* history of low adherence to treatment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women aged 18-90 years with arterial hypertension grade 1-3, stage I-II and initially achieved target BP levels while taking 2-3-component AHT.
Sampling Method: Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2015-09-29 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of BP increasing higher the target level when taking the same therapy | 1-6 months
  Assessment of attenuation of efficacy of previously adequate antihypertensive therapy by using different BP measurement methods

SECONDARY OUTCOMES:
Disease course: assessment of major CVE and death occurrence | 10 years
  Assessment of the disease course depending on the characteristics of 3-6th months of observation

CONTACTS AND LOCATIONS:
Locations (1):
- Oksana Mikhailova, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No